CLINICAL TRIAL: NCT04071691
Title: The PET Imaging of Giant Cell and Takayasu Arteritis Study
Brief Title: PET Imaging of Giant Cell and Takayasu Arteritis
Acronym: PITA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Wellcome Trust (Other); Imperial College London (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Jason Tarkin, Wellcome Clinical Research Career Development Fellow, University of Cambridge
Other Study IDs: A095007 (PITA)
Record Dates: First submitted 2019-08-16; First posted 2019-08-28 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Giant Cell Arteritis; Takayasu Arteritis
MeSH Terms: conditions — Giant Cell Arteritis; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active LVV: Patients with active LVV
  Interventions: Diagnostic Test: PET-MRI
- Stable LVV: Patients with inactive LVV
  Interventions: Diagnostic Test: PET-MRI

INTERVENTIONS:
Diagnostic Test: PET-MRI — SST2 PET-MRI scan

SUMMARY:
While 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) imaging is often included in the diagnostic work-up of patients with large-vessel vasculitis (LVV), 18F-FDG lacks specificity for inflammatory cells and has limited ability to track therapy response. Moreover, high background 18F-FDG uptake in the brain and myocardium largely precludes imaging temporal arteritis in giant-cell arteritis (GCA) and coronary artery involvement in Takayasu arteritis respectively. These limitations of 18F-FDG for imaging LVV highlight important unmet clinical needs, which might be overcome by using a somatostatin receptor subtype-2 (SST2) PET tracer.

DETAILED DESCRIPTION:
Up-regulation of SST2 in activated macrophages represents a novel imaging target for measuring vascular inflammation, which has been previously examined in atherosclerosis using 68Ga-DOTATATE. To test the hypothesis that SST2 PET imaging can accurately identify LVV, patients with active GCA or Takayasu arteritis will undergo vascular 68Ga-DOTATATE or 18F-fluoroethyltriazole-(Tyr3)-octreotate (FETO) PET-MRI at baseline, with repeat imaging after 6 months of treatment. A group of individuals with LVV in clinical remission will also undergo SST2 PET imaging. Data from patients with clinically inactive disease will serve to confirm tracer specificity for active disease, as well as signal reproducibility. 18F-FETO is an alternative SST2 tracer to 68Ga-DOTATATE; the longer half-life and shorter positron range of 18F compared to 68Ga may offer several advantages, including wider tracer availability and improved spatial resolution when imaging small arteries. All patients will also undergo 18F-FDG imaging before treatment, where clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants >18 years old
* Able to give written, informed consent and to lie flat
* Either:

  1. New clinical diagnosis or acute flare of LVV (Giant-cell arteritis or Takayasu's arteritis) within ~1 week of treatment initiation, and
  2. Clinical indication for 18F-FDG PET-CT scan determined by the referring physician, or
  3. Undergoing surgery for LVV, or
  4. Diagnosis of LVV in remission

Exclusion Criteria:

* Women of child bearing potential not using adequate contraception
* Contra-indication to MRI scanning
* Contrast allergy or contrast-nephropathy
* Chronic kidney disease (eGFR <30 mL/min/1.73 m2)
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study
* History of recent malignancy deemed relevant to the study by the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with LVV
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of SST2 PET-MRI for LVV | Baseline
  To determine the diagnostic accuracy of SST2 PET-MRI for LVV, with the clinically adjudicated diagnosis as the gold-standard.

SECONDARY OUTCOMES:
Treatment response | 6 months
  To compare vascular SST2 PET pre- and post-treatment for LVV
Active versus inactive disease | Baseline
  To compare vascular SST2 PET in patients with active disease versus inactive disease
Comparison with biochemical markers of disease severity | Baseline and 6 months
  To compare SST2 PET to C-reactive protein (CRP)
Comparison with clinical measures of disease severity | Baseline and 6 months
  To compare SST2 PET to clinical disease activity scores
Comparison of SST2 PET tracers | Baseline and 6 months
  To compare 68Ga-DOTATATE PET to 18F-FETO PET

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Tarkin, MBBS PhD, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - University of Cambridge, Cambridge, Cambridgeshire
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306
- [Background] Pedersen SF, Sandholt BV, Keller SH, Hansen AE, Clemmensen AE, Sillesen H, Hojgaard L, Ripa RS, Kjaer A. 64Cu-DOTATATE PET/MRI for Detection of Activated Macrophages in Carotid Atherosclerotic Plaques: Studies in Patients Undergoing Endarterectomy. Arterioscler Thromb Vasc Biol. 2015 Jul;35(7):1696-703. doi: 10.1161/ATVBAHA.114.305067. Epub 2015 May 14. PMID 25977567
- [Background] Dubash SR, Keat N, Mapelli P, Twyman F, Carroll L, Kozlowski K, Al-Nahhas A, Saleem A, Huiban M, Janisch R, Frilling A, Sharma R, Aboagye EO. Clinical Translation of a Click-Labeled 18F-Octreotate Radioligand for Imaging Neuroendocrine Tumors. J Nucl Med. 2016 Aug;57(8):1207-13. doi: 10.2967/jnumed.115.169532. Epub 2016 May 12. PMID 27173162